CLINICAL TRIAL: NCT00082160
Title: fMRI Investigation of Meditation
Brief Title: Brain Imaging Technology to Examine the Effects of Meditation
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: K01AT000694-01 (NIH)
Record Dates: First submitted 2004-04-30; First posted 2004-05-04 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Healthy
Keywords: Meditation; Relaxation
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Meditation
Procedure: Functional Magnetic Resonance Imaging

SUMMARY:
The purpose of this study is to use brain imaging technology to identify the parts of the brain that are activated during meditation and to compare these parts to those activated during other activities. This study will also determine the effects of meditation on involuntary functions, such as breathing.

DETAILED DESCRIPTION:
Meditation and relaxation-based interventions are becoming more widely accepted in clinical settings because of their low cost, low risk, and proven effectiveness as a complementary intervention in a wide range of diseases. Despite the success and growing use of relaxation-based treatments, few studies have addressed the basic mechanism by which these treatments work. This study will use functional magnetic resonance imaging (fMRI) to define the brain mechanisms underlying the meditative state, to differentiate this state from other states, and to determine how meditation-induced brain changes affect autonomic function.

Participants in this study will have an fMRI brain scan. Brain activity, breathing rate, and heart rate will be measured while the participant engages in three different activities: lying quietly, meditating, and mentally generating numbers.

ELIGIBILITY:
Inclusion Criteria:

* Daily practice of Vipassana or Kundalini meditation for at least 1 year and participation in at least one 1-week meditation retreat

Exclusion Criteria:

* Current medical or psychological illness
* Use of antidepressants, antianxiolytics, or compounds that alter cerebral blood flow
* Claustrophobia
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2001-07; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital Department of Psychiatry
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States